CLINICAL TRIAL: NCT01126112
Title: Phase II Study of First-line Single-agent Panitumumab in Frail Elderly Patients With Advanced Wild Type K-RAS Colorectal Cancer
Brief Title: Study of First-line Single-agent Panitumumab in Frail Elderly Patients With Advanced Wild Type K-RAS Colorectal Cancer
Acronym: FRAIL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Cooperative Group for the Treatment of Digestive Tumours (TTD) (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TTD-09-03; 2009-016661-28 (EudraCT Number)
Record Dates: First submitted 2010-05-17; First posted 2010-05-19 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Colorectal Cancer
Keywords: advanced colorectal cancer; K-RAS; panitumumab; advanced Wild Type K-RAS colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Panitumumab (Experimental): Panitumumab: 6 mg/Kg Q2W Treatment cycles repeated every 14 days. Subjects will be evaluated for tumour response every 3 cycles (6 wks ± 1 wk) the first 24 weeks and every 8 weeks ± 2 weeks thereafter (per the revised-RECIST 1.1 guideline) until PD or withdrawal from the trial.
  Interventions: Biological: Panitumumab

INTERVENTIONS:
Biological: Panitumumab — Panitumumab: 6 mg/Kg Q2W

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of first-line single-agent panitumumab in frail elderly patients with advanced Wild Type K-RAS colorectal cancer

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the efficacy and safety of first-line single-agent panitumumab in frail elderly patients with advanced Wild Type K-RAS colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

* Signed Inform Consent
* Age > 70 years.
* Histologically documented metastatic colorectal cancer not candidate for surgical resection
* Wild type K-RAS
* Measurable disease by RECIST Criteria
* Intermediate or High-risk group according to the Köhne Prognostic Classification
* ECOG status < 3
* Magnesium ≥ institutional lower limit of normal
* frail elderly patients and or not candidates for chemotherapy:

Frail elderly patients: Presence of one or more of the following criteria:

* Dependence for one of the basic daily living activities (Katz Index)
* Three or more comorbid conditions according Charlson scale and dependence for one of the instrumental activities of daily living (IADL)
* Presence one or more of the following geriatric syndromes (age > 85 years, fecal or urinary incontinence in the absence of stress, frequent falls, spontaneous bone fractures, neglect)

Presence of one or more of the following criteria that make patients not candidates for chemotherapy:

* neutrophils < 2000/mm3
* platelets < 100.000/mm3
* creatinine clearance < 30 ml/min and bilirubin levels > 1.5 x ULN
* creatinine clearance < 30 ml/min and AST or ALT levels > 3 x UNL (if liver metastasis > 5 x ULN)

Exclusion Criteria:

* Patients will be excluded from the study if they have received prior systemic therapy for the treatment of metastatic colorectal carcinoma or antiEGFR therapy, with the exception of adjuvant fluoropyrimidine-based chemotherapy given at least six months prior to enrolment or oxaliplatin at least 12 months prior to enrolment.
* Systemic chemotherapy, hormonal therapy, immunotherapy or experimental or approved proteins/antibodies (eg, bevacizumab) ≤ 30 days before inclusion
* Unresolved toxicities from prior systemic therapy that, in the opinion of the investigator, does not qualify the patient for inclusion
* Patients cognitively impaired or with severe depression according mini mental state examination and geriatric depression scale.
* Patients with central nervous system metastases, or those with significant cardiovascular disease, will also be excluded.
* History of interstitial pneumonitis or pulmonary fibrosis or evidence of interstitial pneumonitis or pulmonary fibrosis on baseline chest CT scan
* Treatment for systemic infection within 14 days before initiating study treatment
* Radiotherapy < 14 days prior to inclusion in the study.
* Active inflammatory bowel disease or other bowel disease causing chronic diarrhoea (defined as > 4 loose stools per day)
* History of any medical condition that may increase the risks associated with study participation or may interfere with the interpretation of the study results
* Known positive test for human immunodeficiency virus infection, hepatitis C virus, chronic active hepatitis B infection
* subject allergic to the ingredients of the study medication or to Staphylococcus protein A
* Any co-morbid disease that would increase risk of toxicity
* Any investigational agent within 30 days before enrolment
* Must not have had a major surgical procedure within 28 days of enrolment
* Subject unwilling or unable to comply with study requirements

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Progression-free survival rate at 6 months | May 2010 - March 2012

SECONDARY OUTCOMES:
Progression-free survival | May 2010 - March 2012
Objective Response Rate | May 2010 - March 2012
Disease control rate | May 2010 - March 2012
Time to response | May 2010 - March 2012
Time to progression | May 2010 - March 2012
Time to treatment failure | May 2010 - March 2012
Duration of response | May 2010 - March 2012
Duration of stable disease | May 2010 - March 2012
Overall survival | May 2010 - March 2012
Changes in patient-reported outcomes | May 2010 - March 2012
Adverse events | May 2010 - March 2012
Evaluation of molecular predictive markers for response. | May 2010 - March 2012

CONTACTS AND LOCATIONS:
Overall Officials: Javier Sastre, Study Chair — Hospital Universitario Clínico San Carlos. Madrid. Spain
Locations (1):
- Spanish Cooperative Group for Gastrointestinal Tumour Therapy, Madrid, Spain

REFERENCES:
- [Derived] Sastre J, Massuti B, Pulido G, Guillen-Ponce C, Benavides M, Manzano JL, Reboredo M, Rivera F, Gravalos C, Safont MJ, Martinez Villacampa M, Llovet P, Dotor E, Diaz-Rubio E, Aranda E; Spanish Cooperative Group for the Treatment of Digestive Tumours TTD. First-line single-agent panitumumab in frail elderly patients with wild-type KRAS metastatic colorectal cancer and poor prognostic factors: A phase II study of the Spanish Cooperative Group for the Treatment of Digestive Tumours. Eur J Cancer. 2015 Jul;51(11):1371-80. doi: 10.1016/j.ejca.2015.04.013. Epub 2015 May 8. PMID 25963019
- See also: Related Info — http://www.ttdgroup.org